CLINICAL TRIAL: NCT02713113
Title: Comparison of Three Different Doses Sugammadex Based on Ideal Body Weight for Reversal of Moderate Rocuronium-induced Neuromuscular Blockade in Laparoscopic Bariatric Surgery.
Brief Title: Efficacy of Low Dose Sugammadex in Reversal of NMB in Laparoscopic Barbaric Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 250
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Bariatric Patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group 1 (Active Comparator): patients were given 1.5 mg / kg. of sugammadex administrated (according to the IBW after T2 of TOF)
  Interventions: Drug: sugammadex reversal of neuromuscular blockade
- group II (Active Comparator): patients were given 2 mg / kg. of sugammadex administrated (according to the IBW after T2 of TOF)
  Interventions: Drug: sugammadex reversal of neuromuscular blockade
- group III (Active Comparator): patients were given 4 mg / kg. of sugammadex administrated (according to the IBW after T2 of TOF)
  Interventions: Drug: sugammadex reversal of neuromuscular blockade

INTERVENTIONS:
Drug: sugammadex reversal of neuromuscular blockade

SUMMARY:
the investigators aimed to compare the efficacy and safety of sugammadex at doses of 1.5, 2, and 4 mg/ kg for the reversal of moderate rocuronium-induced neuromuscular blockade in laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Patients were randomly assigned using a randomization-computer program into three groups according to the dose of sugammadex administrated (according to the IBW after T2 of TOF):

Group I: patients were given 1.5 mg / kg. Group II: patients were given 2 mg / kg. Group III: patients were given 4 mg / kg.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients of both sex (BMI > 40 kg.m-2)
* scheduled for elective laparoscopic bariatric surgery (gastric bypass or sleeve surgery) under general anesthesia using rocuronium for tracheal intubation and maintenance of NMB
* aged between 18 and 60 years and classified as ASA II - III

Exclusion Criteria:

* liver and renal dysfunction,
* disabling neuropsychiatric disorders,
* history of stroke, brain trauma in the last 12 months
* hypersensitivity to anesthetics, history of myocardial infarction, congestive heart failure
* difficult tracheal intubation, and known or suspected disorder affecting NMB.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
sugammadex time following a dose of 1.5 mg / kg of sugammadex according to IBW in comparison to 2, and 4 mg / kg, | 2 hrs

SECONDARY OUTCOMES:
extubation time | 2 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Othman, MD, Study Director — ASSUIT UNVERSITY
Locations (1):
- South Egypt Cancer Instuite, Asyut, Egypt